CLINICAL TRIAL: NCT04311320
Title: A Low-Resource Oxygen Blender Prototype for Use in Modified Bubble CPAP Circuits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00008434
Record Dates: First submitted 2020-03-05; First posted 2020-03-17 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Distress Syndrome; Lower Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-Resource Oxygen Blender (Experimental): This is a single-arm study. All participants will receive respiratory support using the investigational device.
  Interventions: Device: Low-Resource Oxygen Blender

INTERVENTIONS:
Device: Low-Resource Oxygen Blender — The device that is being evaluated is a novel low-cost, high access oxygen blender designed to be used in the World Health Organization bCPAP design. It functions by utilizing the Venturi effect, whereby a narrow jet of one fluid (i.e. oxygen) creates a suction effect and entrains surrounding ambient fluid (i.e. room air) into the jet, effectively creating a mixed solution of both fluids. The cost of materials amounts to approximately 1.40 U.S.D. The average time it takes to build a blender and incorporate it into a bCPAP circuit for a new user is approximately 16 minutes. The materials can all be found in a standard hospital, namely 3cc syringes with rubber stops and a 22 gauge hypodermic needle.

SUMMARY:
Purpose: Using a novel oxygen blender prototype with modified bCPAP to manage children 1 month to 5 years of age hospitalized with respiratory distress due to lower respiratory tract infection (LRTI) in low-resource settings is not associated with clinical failure within 1 hour of use.

Aim: To investigate if this novel oxygen blender is safe to use among children 1 month to 5 years old hospitalized for respiratory distress from lower respiratory tract infections in a low-resource setting.

DETAILED DESCRIPTION:
The study will be a prospective cohort feasibility and safety trial. Patients admitted to Chenla Children's Healthcare who meet eligibility criteria will be asked for consent and then enrolled. Once enrolled, the participant will be treated per hospital protocols and stabilized on bCPAP respiratory support. Once stable for 2 hours, the blender will be incorporated into the bCPAP circuit. At this point, the study nurses will begin recording data for the study as well as providing standard medical care per hospital protocols.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for lung disease and require hospitalization
* Admission diagnosis is lower respiratory tract infection or pneumonia or bronchiolitis (any infectious microbe including bacterial, viral, fungal, parasitic)
* Have respiratory distress on presentation to the hospital (cough or trouble breathing plus at least one of the following: <92% despite low flow oxygen, central cyanosis, tachypnea, chest indrawing, nasal flaring, grunting, head nodding, convulsions, lethargy, inability to breastfeed or drink)
* A bCPAP (electronic) machine is not available to use

Exclusion Criteria:

* History of asthma
* Upper airway obstruction
* Diaphragmatic hernia
* Pneumothorax
* Acute Glasgow Coma score <4
* Cleft Palate
* Cyanotic heart disease
* Bleeding disorders
* Imminent death within 2 hours
* Have had abdominal or thoracic surgery

Ages: 0 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2022-03-26 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility as Measured by Clinical Failure | 1 hour
  The primary outcome of this study is the feasibility of the investigational device as measured by clinical failure within 1 hour of installing the blender in the bubble continuous positive airway pressure (bCPAP) circuit. Clinical failure is defined as the occurrence of any of the following patient events: intubation, death, or transfer for higher level of care, or any 2 of the following events; <85% O2 saturation after 30 min of treatment, new signs of respiratory distress, or partial pressure of carbon dioxide greater than 60 mmHg and pH less than 7.2 in capillary blood gas.
  Outcome will be reported as the percent of participants who experience clinical failure within 1 hour after blender installation.

SECONDARY OUTCOMES:
Oxygen Saturation | Approximately 7 days
  Oxygen saturation will be measured with pulse oximeter every 6 hours for the length of hospital submission. Outcome will be reported as mean of all measurements per patient. Units are percent.
Oxygen Concentration of Outflow | Approximately 7 days
  Oxygen concentration of outflow from nasal cannula will be measured with an oxygen analyzer every 6 hours for the length of hospital submission. Outcome will be reported as mean of all measurements per patient. Units are percent oxygen.
Flow of Oxygen from Tank | Approximately 7 days
  Flow of oxygen from tank will be measured with the gauge on the oxygen canister. Measurements will be recorded every 6 hours for the length of hospital submission. Outcome will be reported as mean of all measurements per patient in units of liters per minute.
Continuous Positive Air Pressure (CPAP) Level | Approximately 7 days
  CPAP level (as displayed on CPAP device) will be recorded every 6 hours for the length of hospital submission. Outcome will be reported as mean of all measurements per patient. This outcome measure is reported in units of cm of H2O.
Bubble Continuous Positive Air Pressure (bCPAP) Maintenance | Approximately 7 days
  bCPAP maintenance is defined as the number of times no bubbling in the water column is noted by study staff indicating the need for maintenance. Need for maintenance will be assessed every 2 hours for the length of hospital stay. Number of incidents per patient will be recorded and outcome will be reported as a mean value of all measurements per patient.
Blender Maintenance | Approximately 7 days
  Blender maintenance is defined as the number of times the blender needs to be repaired or replaced per patient. Need for maintenance will be assessed every 2 hours for the length of hospital stay. Number of incidents per patient will be recorded and outcome will be reported as mean value of all measurements per patient.
Duration of Respiratory Support | Approximately 7 days
  Outcome will be reported as the length of time (in hours) that respiratory support (i.e. requiring bCPAP and blender) is required during hospital submission.
Number of Patient Transfers | Approximately 7 days
  Outcome is reported as number of patients who require transfer to a higher level of care.
Number of Patient Intubations | Approximately 7 days
  Outcome is reported as number of patients requiring intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wu, MD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- Chenla Children's Healthcare, Kratié, Kratié Province, Cambodia